CLINICAL TRIAL: NCT01265082
Title: Explore the Mechanisms of Pruritus in Bullous Pemphigoid Patients During Remission
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Li-Fang, Wang, Department of Dermatology, National Taiwan University Hospital
Other Study IDs: 201006012R
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Bullous Pemphigoid; Pruritus
MeSH Terms: conditions — Pemphigoid, Bullous; Pruritus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients in remission with pruritus
- Patients in remission without pruritus

SUMMARY:
The following is the investigators hypothesis regarding the pruritus of BP patients during remission. Anti-BP 180 IgE binds to dermal mast cells, inducing their activation and secretion of mediators after being cross-linked by antigens. Among mediators, histamine directly induces itching and vessel changes, whereas tryptase potentiates itching and vessel changes in an indirect way through the actions of neuropeptides. Tryptase stimulates neurons which in turn secrete neuropeptides.

DETAILED DESCRIPTION:
Bullous pemphigoid(BP) is a cutaneous autoimmune blister disease. In addition to blisters formation which disrupt skin barrier and result in high mortality, erythematous edematous plaques often develop on skin of bullous pemphigoid patients accompanied with intensive pruritus. As regard with the pathogenesis of BP, it is generally accepted that anti-BP180 IgG is the most important pathogenic factor for blister formation, whereas anti-BP180 IgE which binds to mast cells and induces their activation results in erythematous edematous plaques. Quite a few bullous pemphigoid patients suffer from intensive pruritus even during clinical remission period that means blisters or plaques are no longer on their skin. The reasons why pruritus persists during this period are still obscure.

Pruritus is the most common symptom of cutaneous diseases. Our understanding regarding pathophysiology of "pruritus" has made a remarkable progress in the past decade. Now, it is known that there are various kinds of substances that induce pruritus (pruritus mediators) and different combinations of these mediators are involved in different itching diseases. Moreover, neuropeptides secreted by stimulated neurons can in turn induce neurogenic inflammation.

The following is our hypothesis regarding the pruritus of BP patients during remission. Anti-BP 180 IgE binds to dermal mast cells, inducing their activation and secretion of mediators after being cross-linked by antigens. Among mediators, histamine directly induces itching and vessel changes, whereas tryptase potentiates itching and vessel changes in an indirect way through the actions of neuropeptides. Tryptase stimulates neurons which in turn secrete neuropeptides.

Thus, in order to test our hypothesis, the strategy of this study is to compare parameters between two groups of patients, bullous pemphigoid patients in remission with pruritus and without pruritus. The following parameters in serum and skin will be measured: total IgE, anti-BP 180 IgE, the number and activated status of mast cells, the amount of some mediators and neuropeptides produced by mast cells and neurons, respectively. In addition, these parameters in active stage will also be measured for reference and with a hope to find useful parameters for predicting the persistence of pruritus in remission.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bullous pemphigoid

Exclusion Criteria:

* Patients have other disorders which can lead to itching sensation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic,
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsu Cho, M.D., Study Director — Department of Dermatology, National Taiwan University Hospital
Locations (1):
- Department of Dermatology, National Taiwan University Hospital, Taipei, Taiwan